CLINICAL TRIAL: NCT04280783
Title: Feasibility and Acceptability of a Web-based Physical Activity for the Heart (PATH) Intervention Designed to Reduce the Risk of Heart Disease Among Inactive African Americans
Brief Title: Active You: A Novel Exercise Program for African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Jacob Kariuki, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY19110217; 5UL1TR001857-04 (NIH)
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Risk Factor; Prediabetes; Overweight and Obesity; Sedentary Behavior
Keywords: Physical activity; Web-based; YouTube; Remote
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity; Sedentary Behavior; Motor Activity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: We will randomize 30 participants to either the PATH treatment group or wait-list control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PATH Treatment Group (Experimental): The PATH group will be granted password protected access to one of the 3 PATH levels based on their baseline fitness status. The intervention is designed to help participants increase their baseline PA via health coaching, self-monitoring and pragmatic workout videos that provide convenient options for overcoming socio-environmental barriers to PA.
  Interventions: Behavioral: The Physical Activity for The Heart (PATH) intervention
- Wait-list control group (Other): Participants in this group will not have access to the PATH intervention until after 12 weeks when they cross over. After randomization, the control group will be provided with a copy of the Be Active Your Way booklet, developed by the Centers for Disease Control (CDC) to help individuals integrate PA in their daily lives.
  Interventions: Behavioral: Be Active Your Way Booklet

INTERVENTIONS:
Behavioral: The Physical Activity for The Heart (PATH) intervention — The web-based Physical Activity for The Heart (PATH) intervention leverages openly accessible platforms, such as YouTube, to proffer workout videos that match the participants preferences. Currently, PATH includes over 90 workout videos vetted by a team of experts and curated on the PATH website in 3 controlled levels of intensity (beginner, intermediate, proficient) to foster gradual progression from low to high intensity PA in accordance with the FITT-VP (frequency, intensity, time, type, volume, progression) principle.
  Arms: PATH Treatment Group
Behavioral: Be Active Your Way Booklet — Be Active Your Way booklet was developed by the Centers for Disease Control (CDC) to help individuals integrate PA in their daily lives. It simply encourages individuals to increase their PA gradually and gives them examples of things that they can do.
  Arms: Wait-list control group

SUMMARY:
Barriers to physical activity (PA) among African Americans (AAs) have been extensively studied, yet there is a paucity of innovative PA interventions designed to address them. In recent years, many studies have used the internet to promote PA in many settings, including the home environment, but only a few studies have recruited AAs. Without innovative and culturally relevant interventions, AAs will continue reporting extremely low levels of PA and disparate cardiovascular health outcomes. In prior work, the investigators sought the input of AA focus groups to inform the development of a technology-based Physical Activity for The Heart (PATH) intervention that leverages openly accessible platforms, such as YouTube, to promote PA in any setting. The investigators designed PATH as a culturally salient action-oriented intervention that can be accessed in any setting to promote PA among inactive AAs. In this application, the investigators propose to examine whether PATH is a feasible strategy for promoting PA among inactive AAs. In Aim 1 the investigators will conduct a randomized clinical trial that will include 30 inactive AAs to assess the feasibility and acceptability of the PATH intervention. In Aim 2 the investigators will examine the trend in PA and cardiovascular disease risk change from baseline to post-intervention. This approach is innovative because it leverages openly accessible technologies to provide a wide variety of free, enjoyable and action-oriented workout videos that match AAs preferences. This contribution will be significant because PATH could offer a novel, low-cost, and scalable strategy for promoting PA among individuals facing socio-environmental barriers to PA.

DETAILED DESCRIPTION:
Whereas an inverse dose-response relationship has been established between physical activity (PA) and a host of chronic illnesses, including cardiovascular disease (CVD), most American adults (79%) are physically inactive and do not attain the minimum PA levels recommended by the PA Guidelines for Americans. African Americans (AAs) in particular report very low levels of PA, and have the highest burden of CVD in the United States.To eliminate the prevailing cardiovascular health disparities, there is a critical need for pragmatic and culturally salient interventions that are designed to address barriers to PA that are more problematic for AAs.

Common barriers to PA such as lack of time and low exercise self-efficacy are pervasive in all racial groups. In addition to these barriers, socio-environmental factors, such as unsafe neighborhoods and limited access to fitness facilities play a key role in perpetuating the low levels of PA observed in AAs. To mitigate these barriers, home-based PA interventions delivered via mail, telephone and internet have been developed. Although only a few of these interventions have been tested among AAs, preliminary studies have reported more participation and retention of AAs in home-based PA programs. However, the associated PA outcomes have been minimal, especially in less educated AAs. Low literacy levels and reliance on print-based resources with no cultural appeal are thought to limit the utility of the interventions in AAs. The investigators have previously reported how AAs prefer PA programs that are visual, convenient, fun to engage in, and feature people they can relate to especially in body size, fitness status and age. Other studies have reported similar preferences for PA among AAs, yet there is a paucity of PA interventions that are designed to incorporate these preferences.

To bridge this gap, the investigators have developed a web-based Physical Activity for The Heart (PATH) intervention that leverages openly accessible platforms, such as YouTube, to proffer workout videos that match the reported preferences. Currently, PATH includes 90 workout videos vetted using the FITT principle (frequency, intensity, time, type) and curated on the PATH website in 3 controlled levels of intensity (beginner, intermediate, proficient) to foster gradual progression from low to high intensity PA. The overarching aim of the proposed study is to conduct a pilot randomized controlled trial (RCT) to assess the feasibility and acceptability of the PATH intervention for promoting PA in AAs. The investigators will enroll 30 inactive AAs and randomize them to either treatment (12-wks of PATH) or wait-list control (use a general health handout) group to address the following specific aims:

Aim 1: Assess the feasibility and acceptability of the PATH intervention among inactive AAs. Feasibility will be assessed via 1) number of participants screened for eligibility; 2) percentage eligible; 3) percentage enrolled; 4) percentage retained within each randomized group; and 5) adherence to self-monitoring (Actigraph wear time) and intervention protocol (PATH utilization). Acceptability will be evaluated via a post-intervention survey developed by the study team to appraise the intervention's usability and perceived efficacy for increasing PA.

Aim 2: Describe the trends in PA and CVD risk change from baseline to post-intervention. The primary outcome will be PA and will include objectively measured steps, light PA, and moderate-to-vigorous PA (MVPA). Cardiovascular outcomes will include blood pressure (BP), body fat percentage, body mass index (BMI), glycated hemoglobin (HbA1c) and lipids (LDL, HDL, and total cholesterol). Trends will be summarized as mean within-group changes (with 95% confidence intervals [CIs]).

The proposed research addresses a key driver of cardiovascular health disparities and is innovative in its rigorous testing of the novel PATH intervention for feasibility and acceptability among inactive AAs. Findings from this study will inform the refinement of the PATH intervention to be tested in a full-scale RCT.

ELIGIBILITY:
Inclusion Criteria:

1. 40-70 years old
2. BMI≥25
3. Have regular access to the internet (via computer or smart phone)
4. Less than 90 mins of self-reported moderate to vigorous physical activity per week
5. American Diabetes Association (ADA) risk ≥5
6. Available for pre and post-intervention assessments.
7. Self-identify as Black/African American

Exclusion Criteria:

1. Unstable conditions that may require supervised PA
2. Physical limitations that may prohibit engagement in MVPA
3. Pregnancy or intention to become pregnant during study, history of CVD
4. Current participation in a PA study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Kariuki, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Primay Health Network, Beaver Falls, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
It is our goal to make all data generated from this proposal available to other investigators without compromising the confidentiality of participants. Investigators who would like to do a secondary analysis of de-identified data can submit a formal request for the data including the proposal of their intended analysis to the PI at activeu@pitt.edu. The PI will review all requests and facilitate data access once approval is granted.
Supporting Information: SAP, CSR
Time Frame: 12 months after the end of the study
Access Criteria: Data access will be provided based on scientific merit of the proposed analysis, IRB approval and data agreement contract as deemed appropriate by University of Pittsburgh

REFERENCES:
- [Derived] Kariuki JK, Sereika S, Erickson K, Burke LE, Kriska A, Cheng J, Milton H, Hirshfield S, Ogutu D, Gibbs B. Feasibility and preliminary efficacy of a novel web-based physical activity intervention in adults with overweight/obesity: A pilot randomized controlled trial. Contemp Clin Trials. 2023 Oct;133:107318. doi: 10.1016/j.cct.2023.107318. Epub 2023 Aug 23. PMID 37625586

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PATH Treatment Group | Wait-list Control Group
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1
Not completed — Family issues unrelated to the study. | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Wait-list Control Group: Participants in this group will not have access to the PATH intervention until after 12 weeks when they cross over. After randomization, the control group will be provided with a copy of the Be Active Your Way booklet, developed by the Centers for Disease Control (CDC) to help individuals integrate PA in their daily lives.
  Be Active Your Way Booklet: Be Active Your Way booklet was developed by the Centers for Disease Control (CDC) to help individuals integrate PA into their daily lives. It simply encourages individuals to increase their PA gradually and gives them examples of things that they can do.
- Total: Total of all reporting groups
Arm/Group | PATH Treatment Group | Wait-list Control Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (8.0) | 55.9 (8.5) | 55.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 15 | 15 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Body Mass Index [Mean (Standard Deviation); unit: Kg/M^2] | 38.29 (7.56) | 37.08 (6.63) | 37.69 (7.01)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 120.33 (17.37) | 124.07 (19.50) | 122.20 (18.24)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 79.87 (10.11) | 81.50 (10.66) | 80.68 (10.24)
Objective weekly MVPA minutes [Mean (Standard Deviation); unit: Minutes] — Objective Moderate to Vigorous Physical Activity (MVPA) was measured using waist-worn Actigraph GT3X. Freedson Adult (1998) cutpoints were used.
  Minutes | 169.73 (159.86) | 156.60 (127.53) | 163.17 (142.25)
Adherence to MVPA guidelines at baseline [Number; unit: participants] — This measure describes the proportion of the sample that met the recommended minimum physical activity levels (150 MVPA minutes) at baseline.
  participants | 5 | 5 | 10
Objective average daily steps [Mean (Standard Deviation); unit: Steps] | 2923.6 (2897.4) | 1983.11 (2418.76) | 2910.5 (2173.26)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Retained at the End of Study
Description: Will be indicated by the number of enrolled participants who are retained by the end of the study.
Time Frame: Post-intervention at 12 weeks
Population: All participants enrolled in the study
Measure: Number; unit: Percent of enrolled participants
Arm/Group | PATH Treatment Group | Wait-list Control Group
Number analyzed (Participants) | 15 | 15
Percent of enrolled participants | 93.33 | 93.33

2. Primary Outcome: Percentage of Participants Who Self-monitored Step Count Using Wrist Worn ActiGraph GT9X Over the Study Period
Description: will be indicated by the proportion of the sample with ≥4days per week of valid Actigraph wear time (≥10hrs) during the entire course of the study.
Time Frame: Post-intervention at 12 weeks
Measure: Number; unit: percentage of the sample
Arm/Group | PATH Treatment Group | Wait-list Control Group
Number analyzed (Participants) | 14 | 14
percentage of the sample | 92.86 | 71.43

3. Primary Outcome: Acceptability of PATH Intervention
Description: Percentage of participants who reported the PATH platform was culturally appropriate
Time Frame: Post-intervention at 12 weeks
Measure: Number; unit: percentage of intervention participants
Arm/Group | PATH Treatment Group | Wait-list Control Group
Number analyzed (Participants) | 14 | 14
percentage of intervention participants | 100 | 92.86

4. Secondary Outcome: Body Mass Index (BMI) at 12 Weeks
Description: BMI will be measured using Fitbit Aria II scale provided to the participant by the study team. The study team will guide the participants on how to measure their BMI and will supervise the measurement via HIPAA compliant Zoom session.
Time Frame: Post-intervention at 12 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | PATH Treatment Group | Wait-list Control Group
Number analyzed (Participants) | 14 | 14
kg/m^2 | 37.62 (7.85) | 36.65 (6.43)

5. Secondary Outcome: Change From Baseline in Body Fat Percentage at 12 Weeks
Description: Body fat percentage will be measured using Fitbit Aria II scale provided to the participant by the study team. The study team will guide the participants on how to measure their body fat and will supervise the measurement via HIPAA compliant Zoom session.
Time Frame: Post-intervention at 12 weeks
Measure: Mean (Standard Error); unit: body fat percentage
Arm/Group | PATH Treatment Group | Wait-list Control Group
Number analyzed (Participants) | 13 | 14
body fat percentage | -1.445 (.377) | -.522 (.426)

6. Secondary Outcome: Change From Baseline in Waist Circumference at 12 Weeks
Description: Waist circumference will be measured using Perfect waist tape measure provided to the participant by the study team. The study team will guide the participants on how to take the measurement using a standard video and will be able to observe the outcome of the measurement via HIPAA compliant Zoom session.
Time Frame: Post-intervention at 12 weeks
Measure: Mean (Standard Error); unit: Inches
Arm/Group | PATH Treatment Group | Wait-list Control Group
Number analyzed (Participants) | 14 | 14
Inches | -.182 (.793) | -.948 (.499)

7. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at 12 Weeks
Description: Both diastolic and systolic BP will be reported. The measurement will be done using automated OMRON BP machine provided to the participant by the study team. The study team will guide the participants on how to take blood pressure and will supervise the measurement via HIPAA compliant Zoom session.
Time Frame: Post-intervention at 12 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | PATH Treatment Group | Wait-list Control Group
Number analyzed (Participants) | 14 | 14
mmHg | -1.869 (4.107) | -3.899 (3.744)

8. Secondary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1C) at 12 Weeks
Description: The sample for HbA1C will be collected by participants at home using the dry blood spot method. The study team will guide the participants on how to take the sample using a standard video and will supervise the collection via HIPAA compliant Zoom session. The sample will be processed by CoreMedica lab using standard protocols
Time Frame: Post-intervention at 12 weeks
Measure: Mean (Standard Error); unit: Percentage of glycated hemoglobin"
Arm/Group | PATH Treatment Group | Wait-list Control Group
Number analyzed (Participants) | 9 | 10
Percentage of glycated hemoglobin" | .007 (.118) | .072 (.112)

9. Secondary Outcome: Change From Baseline in Total Cholesterol at 12 Weeks
Description: The blood sample for lipids (total cholesterol) will be collected by participants at home using the dry blood spot method. The study team will guide the participants on how to take the sample using a standard video and will supervise the collection via HIPAA compliant Zoom session. The sample will be processed by CoreMedica lab using standard protocols.
Time Frame: Post-intervention at 12 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | PATH Treatment Group | Wait-list Control Group
Number analyzed (Participants) | 10 | 9
mg/dL | 10.623 (12.932) | -13.363 (12.281)

10. Secondary Outcome: Change From Baseline in the Risk Score for Diabetes at 12 Weeks
Description: The risk score for diabetes will be measured via the American Diabetes Association (ADA) Risk Calculator. The scores range from 0 to 10 with higher scores indicating high risk for developing type 2 diabetes.
Time Frame: Post-intervention at 12 weeks
Population: End of study ADA score data were not collected
Arm/Group | PATH Treatment Group | Wait-list Control Group
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in Step Count at 12 Weeks
Description: Step count will be measured using a wrist worn ActiGraph GT9X link during the entire study period. The study outcomes will focus on change from baseline to 12 weeks
Time Frame: Post-intervention at 12 weeks
Measure: Mean (Standard Error); unit: Steps
Arm/Group | PATH Treatment Group | Wait-list Control Group
Number analyzed (Participants) | 14 | 14
Steps | 618.633 (235.36) | 239.965 (401.713)

12. Secondary Outcome: Moderate to Vigorous Physical Activity
Description: Change from baseline in moderate to vigorous physical activity (MVPA) at 12 weeks measured using a waist worn ActiGraph GT3X accelerometer
Time Frame: Post-intervention at 12 weeks
Measure: Mean (Standard Error); unit: Minutes
Arm/Group | PATH Treatment Group | Wait-list Control Group
Number analyzed (Participants) | 14 | 14
Minutes | 33.498 (22.025) | 18.582 (26.221)

13. Secondary Outcome: Change From Baseline in Barriers Exercise Self-efficacy (BARSE) Scale at 12 Weeks
Description: Participants will be asked to respond to the BARSE scale appraising their exercise self-efficacy. The scale range from 0 to 100, with higher scores indicating increased exercise self-efficacy
Time Frame: Post-intervention at 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PATH Treatment Group | Wait-list Control Group
Number analyzed (Participants) | 14 | 14
score on a scale | 54.4 (6.5) | 56.9 (6.4)

14. Other Pre Specified Outcome: Change From Baseline in Light Physical Activity at 12 Weeks
Description: Light physical activity will be measured using a waist worn ActiGraph GT3X accelerometer
Time Frame: Post-intervention at 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The adverse events data was collected over 12 weeks for intervention group and 24 weeks for control group (because they crossed over to use the intervention after 12 weeks).
Arm/Group | PATH Treatment Group | Wait-list Control Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
The short study length and small sample size limit our ability to test effectiveness; however, as our study was meant to demonstrate feasibility and acceptability, in line with the ORBIT model, this is appropriate for the formative phase of behavioral intervention development.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT04280783/Prot_001.pdf
  • Informed Consent Form (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT04280783/ICF_000.pdf